CLINICAL TRIAL: NCT01240096
Title: Phase 4 Study of Mirtazapine in Functional Dyspepsia Patients With Weight Loss
Brief Title: Mirtazapine Versus Placebo in Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Jan Tack, M.D., Ph.D., University Hospitals Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S50181
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Functional Dyspepsia
Keywords: Functional dyspepsia; Weight loss; Mirtazapine
MeSH Terms: conditions — Weight Loss | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirtazapine (Active Comparator): mirtazapine 15 mg daily
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine 15 mg daily
  Other Names: mirtazapine is Remergon

SUMMARY:
Double-blind randomized controlled trials of 8 weeks mirtazapine 15 mg daily or placebo, followed by 8 weeks of open-label mirtazapine 15 mg daily

DETAILED DESCRIPTION:
Double-blind randomized controlled trials of 8 weeks mirtazapine 15 mg or placebo, followed by 8 weeks of open-label mirtazapine

Two weeks run-in, 8 weeks randomized, 8 weeks open label

Assessments include

* dyspepsia questionnaire
* Nepean dyspepsia index
* Daily diary
* Vital signs

ELIGIBILITY:
Inclusion Criteria:

* Functional dyspepsia according to Rome II criteria
* Weight loss of > 5% body weights

Exclusion Criteria:

* Organic GI pathology
* History of upper gi tract surgery
* Major depression or anxiety
* Use of antidepressants in the last 2 months
* Prokinetic drugs or spasmolytic drugs
* Analgesic use (except paracetamol)
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2012-09-11 (Actual)

PRIMARY OUTCOMES:
Difference in dyspepsia symptom scores week 8 versus week 0 | Week 8 compared to week 0
  The Dyspepsia Symptom Score is calculated from the dyspepsia symptom severity questionnaire at weeks 0, 4 and 8. The symptom score has been used in previous studies (Tack et al., Gastroenterology 1998).

SECONDARY OUTCOMES:
Individual symptom severities | Week 8 compared to week 0
  Individual symptom scores from the dyspepsia symptom score (DSS) which is used as primary endpoint
Nepean dyspepsia index for quality of life in functional dyspepsia | Week 8 compared to week 0
  Use of the validated NDI.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals, Leuven, Flanders, Belgium

REFERENCES:
- [Derived] Tack J, Ly HG, Carbone F, Vanheel H, Vanuytsel T, Holvoet L, Boeckxstaens G, Caenepeel P, Arts J, Van Oudenhove L. Efficacy of Mirtazapine in Patients With Functional Dyspepsia and Weight Loss. Clin Gastroenterol Hepatol. 2016 Mar;14(3):385-392.e4. doi: 10.1016/j.cgh.2015.09.043. Epub 2015 Oct 30. PMID 26538208
- See also: Website Research Group — http://www.targid.eu